CLINICAL TRIAL: NCT02586389
Title: Collection of Whole Blood and Tissue Specimens from Patients Diagnosed with Non-Hematologic Cancer for Use in Development of a Noninvasive Liquid Biopsy Assay to Determine the Tumor Genomic Profile in Circulating Cell-Free Tumor DNA
Brief Title: Specimen Collection from Patients with Non-Hematologic Cancer for Use in Development of a Liquid Biopsy Assay
Status: Recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-CA-101
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Non-hematologic Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and tissue samples will be collected for DNA extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-hematological Cancer Cohort: Eligible subjects will have been previously diagnosed with a non-hematological cancer with tumor present at baseline blood draw.

SUMMARY:
This specimen collection is designed to obtain whole blood and tumor tissue from subjects diagnosed with cancer for the purpose of the development of a noninvasive liquid biopsy assay using next generation sequencing (NGS).

DETAILED DESCRIPTION:
This is a non-significant risk multicenter, longitudinal specimen collection study. At the Baseline Visit, whole blood will be collected to be paired with either a previously collected tumor biopsy tissue sample or a prospectively collected tumor tissue sample. Whole blood samples will also be collected longitudinally at Interim visits for up to 5 years. Interim visits will be on a schedule dictated by their physician's standard-of-care management protocol. No more than 100mL of blood will be collected per month. Tumor tissue from recurrences will be collected for the duration of subject participation (after the Baseline Visit).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older;
* Subject is willing to provide written informed consent;
* Subject has a diagnosis of a non-hematologic cancer, has tumor in the body, and has either;

  1. residual tumor tissue available for testing by the Sponsor; or
  2. genomic profiling results from an IVD or LDT assay performed on tumor biopsy tissue; or
  3. an invasive procedure (biopsy, surgery) scheduled following the Baseline Visit from which residual tumor tissue can be available for testing by the Sponsor.
* Subject is able, in the professional opinion of the investigator, to provide whole blood at the Baseline Visit and at the Interim Visits.

Exclusion Criteria:

* Underwent curative-intent surgery for management of the presently diagnosed tumor, at any time prior to the Baseline Visit.
* Underwent targeted or non-targeted chemotherapy, hormone receptor blocking therapy, or radiation therapy prior to the Baseline Visit.
* Underwent an invasive procedure (biopsy, surgery, thermal ablation) in the 7 days prior to any blood collection (baseline or follow-up).
* Any medical or mental condition that would interfere with the subjects' ability to willingly give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients at least 18 years of age who have been diagnosed with non-hematologic cancer (Stages I-IV) and who meet all study inclusion criteria and no exclusion criteria. Primarily subjects with breast, colorectal, lung, or melanoma cancer (90%) will be enrolled. The remaining subjects (10%) diagnosed with other cancer types may be enrolled on a case by case basis.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-10-13 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
biospecimen sample collection for liquid biopsy assay development | After cancer diagnosis through 5 years of standard of care follow-up visits
  Analysis of circulating tumor DNA (ctDNA) in whole blood will be compared to baseline tumor DNA for concordance of mutations related to cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Beruti, MD, Study Director — Sequenom, Inc.
Locations (1):
- Idaho Urology, Boise, Idaho, United States